CLINICAL TRIAL: NCT06663358
Title: A Multi-Country Observational Study of Safety and Effectiveness of Elfabrio® in Fabry Patients
Acronym: MODERN
Status: Recruiting | Type: Observational
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLI-06657AA1-10
Record Dates: First submitted 2024-09-23; First posted 2024-10-29 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2024-11

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cardiac Cohort: Patients with Fabry-related cardiac disease
  Interventions: Drug: Pegunigalsidase-alfa
- Naïve Cohort: Patients naïve to prior Fabry disease treatment
  Interventions: Drug: Pegunigalsidase-alfa
- Long-Term Cohort: Patients previously participating in the pegunigalsidase alfa open label extension study and transitioning to routine care
  Interventions: Drug: Pegunigalsidase-alfa

INTERVENTIONS:
Drug: Pegunigalsidase-alfa — Administered via intravenous (IV) infusion under conditions of routine clinical care
  Other Names: Elfabrio®

SUMMARY:
A multi-centre, multi-country, observational, non-interventional, retrospective and prospective (hybrid) study among Fabry disease participants treated with pegunigalsidase alfa (Elfabrio®) in routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged > 18 years of age at the time of consent.
* Genetically confirmed diagnosis of Fabry disease.
* Either taking or planning to take pegunigalsidase alfa as treatment for Fabry disease.
* No contraindications for cardiac magnetic resonance imaging (cMRI)
* Informed consent form (ICF) signed and dated indicating the individual has been informed of and agreed to all pertinent aspects of the study and is willing to comply with all study requirements, including completion of electronic patient reported outcomes (ePROs).
* Cardiac Cohort:
* Evidence of Fabry disease (FD)-related heart disease including one or more of the following:
* Left ventricular hypertrophy (LVH) measured by left ventricular mass index (LVMI) (g/m2) elevation above age/sex specific reference ranges.
* Posterior septum wall thickness (e.g., >=13mm) not explained by other factors (e.g., hypertension)
* Low native T1 mapping on cMRI.
* Typical Fabry-like scar on cMRI
* Participants can receive cardiac magnetic resonance imaging (cMRI) with gadolinium enhancement as part of their SoC.
* Estimated glomerular filtration rate (eGFR) >45 mL/min/1.73 m2, assessed within the prior 6 months.
* Naïve Cohort:
* Most recent eGFR>45 mL/min/1.73 m2, assessed within prior 6 months.
* Male participants should have abnormal elevation in plasma lysoGb3 as assessed within 6 months prior to enrolment.
* Long-Term Cohort:
* Participants previously enrolled in the open label study CLI-06657AA1-04 (Previously PB-102-F60) (using pegunigalsidase alfa at a dose of 1mg/kg every 2 weeks) who have initiated or plan to initiate commercial pegunigalsidase alfa (Elfabrio®).

Exclusion Criteria:

* Contraindication to magnetic resonance imaging (MRI) including known history of hypersensitivity to gadolinium contrast agent that is not managed by the use of premedication.
* Pregnant at the time of enrolment.
* Presence of any medical, emotional, behavioural, or psychological condition that, in the judgment of the physician, could interfere with the ability to participate in the study.
* Active participation in any interventional study for Fabry disease
* Treatment regimen at the time of enrolment in the study is different from the approved 1mg/kg every two weeks (note if regimen subsequently changes during the prospective part of the study, the participants can remain in the study)
* Prior participation in a pegunigalsidase alfa trial using a dose of 2 mg/kg administered every 4 weeks.
* Cardiac Cohort:
* History of acute myocardial infarction or congestive heart failure with reduced left ventricular (LV) ejection fraction of less than 35%.
* Cerebral vascular accident (CVA) in the prior 6 months.
* Chronic liver cirrhosis.
* FD-unrelated heart disease (e.g., scarring due to myocardial infarction, symptomatic occlusive coronary artery disease, moderate valvular heart disease not thought to be Fabry related).
* The participant is or has been treated with any investigational drug for Fabry disease within 6 months of study start or investigational gene therapy for Fabry disease at any time point in the past.
* Severe cardiac fibrosis defined as more than 3 segments that each have >50% fibrosis upon late gadolinium enhancement cMRI at any prior cMRI.
* Naïve Cohort:
* Prior exposure to a FD therapy (Replagal®, Fabrazyme®, and Galafold®) at any time point.
* Severe cardiac fibrosis defined as more than 3 segments that each have >50% fibrosis upon late gadolinium enhancement cMRI on any prior cMRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The eligible population for this study includes participants who have a genetically confirmed diagnosis of Fabry disease and are being treated or plan to initiate treatment with pegunigalsidase alfa (Elfabrio®). Participants will be required to meet inclusion, not meet exclusion criteria and sign informed consent to be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Estimated Glomerular Filtration Rate (eGFR) | 4 years
  eGFR, calculated using the Chronic Kidney Disease - Epidemiology Collaboration (eGFRCKD-EPI) equation from study baseline and from pegunigalsidase alfa treatment start to end of follow-up and to pre-specified time points (annually).
Plasma Globotriaosylsphingosine (LysoGb3) Concentration | 4 years
  Levels of the Fabry disease biomarker plasma globotriaosylsphingosine (lyso-Gb3) over time, and change from study baseline and from pegunigalsidase alfa treatment start to end of follow-up.
Left Ventricular Mass Index (LVMI; g/m2) | 4 years
  Change in LVMI over time as assessed by cardiac MRI. Based on LVM indexed by height and/or body surface area.
High Sensitivity Troponin (hs-cTnT) | 4 years
  Change in levels of hs-cTnT over time
Safety Assessments | 4 years
  The endpoints will include occurrence of SAEs, infusion-related reactions (IRRs), drug-related adverse events, and proportion of participants with ADAs over time.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Emory University School of Medicine, Atlanta, Georgia
  - Northwestern University - Feinberg School of Medicine - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Infusion Associates, Grand Rapids, Michigan
  - Lysosomal & Rare Disorder Research & Treatment Center (LRDRTC), Fairfax, Virginia
- General Hospital Slovenj Gradec, Slovenj Gradec, Slovenia
- United Kingdom (3):
  - University Hospitals Birmingham NHS Foundation Trust, Queen Elizabeth Hospital, Edgbaston, Birmingham
  - Salford Royal, Salford, Greater Manchester
  - The Royal Free Hospital, London